CLINICAL TRIAL: NCT02913703
Title: Effect of Preprandial Ghrelin on Postprandial Glucose Tolerance
Brief Title: Preprandial Ghrelin Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jenny Tong, MD, MPH (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Jenny Tong, MD, MPH, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00071271; R01DK097550 (NIH)
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes
Keywords: Ghrelin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ghrelin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Healthy subjects - Preprandial AG (Acyl Ghrelin) (Experimental): Control group of healthy subjects. Subjects will eat standardized, provided breakfast at home; then after a 4 hour fast, they will receive a preprandial AG (Acyl Ghrelin) bolus over 1 minute. Sixty minutes later, they will receive a liquid mixed meal (Ensure: 2 cans/474 ml). Venous blood samples will be taken over the entire 245 minutes.
  Interventions: Drug: Ghrelin
- Healthy subjects - Preprandial saline (Experimental): Control group of healthy subjects. Subjects will eat standardized, provided breakfast at home; then after a 4 hour fast, they will receive a preprandial saline bolus over 1 minute. Sixty minutes later, they will receive a liquid mixed meal (Ensure: 2 cans/474 ml). Venous blood samples will be taken over the entire 245 minutes.
  Interventions: Other: Saline
- Healthy subjects - Prandial AG (Experimental): Control group of healthy subjects. Subjects will eat standardized, provided breakfast at home; then after a 5 hour fast, they will receive a prandial AG bolus over 1 minute starting at the same time as the liquid mixed meal (Ensure: 2 cans/474 ml). Venous blood samples will be taken over the entire 245 minutes.
  Interventions: Drug: Ghrelin
- Healthy subjects - Preprandial & prandial AG (Experimental): Control group of healthy subjects. Subjects will eat standardized, provided breakfast at home; then after a 4 hour fast, they will receive a preprandial AG bolus over 1 minute. Sixty minutes later, they will receive another AG bolus over 1 minute starting at the same time as the liquid mixed meal (Ensure: 2 cans/474 ml). Venous blood samples will be taken over the entire 245 minutes.
  Interventions: Drug: Ghrelin
- Diabetic subjects - Preprandial AG (Experimental): Type 2 diabetic subjects will eat standardized, provided breakfast at home; then after a 4 hour fast, they will receive a preprandial AG bolus over 1 minute. Sixty minutes later, they will receive a liquid mixed meal (Ensure: 2 cans/474 ml). Venous blood samples will be taken over the entire 245 minutes.
  Interventions: Drug: Ghrelin
- Diabetic subjects - Preprandial Saline (Experimental): Type 2 diabetic subjects will eat standardized, provided breakfast at home; then after a 4 hour fast, they will receive a preprandial saline bolus over 1 minute. Sixty minutes later, they will receive a liquid mixed meal (Ensure: 2 cans/474 ml). Venous blood samples will be taken over the entire 245 minutes.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Ghrelin — Boluses of Ghrelin will be given over a 1 minute period at 3 ug/kg. Ensure (2 cans) will also be given.
  Arms: Diabetic subjects - Preprandial AG; Healthy subjects - Prandial AG; Healthy subjects - Preprandial & prandial AG; Healthy subjects - Preprandial AG (Acyl Ghrelin)
Other: Saline — Boluses of saline will be given over a 1 minute period. Ensure (2 cans) will also be given.
  Arms: Diabetic subjects - Preprandial Saline; Healthy subjects - Preprandial saline

SUMMARY:
Background and Significance: The peptide hormone ghrelin drives hunger and feeding behavior, making it a focus of obesity research. Released mainly by the stomach and proximal small intestine, ghrelin peaks prior to meals, potentially priming the gut for anticipated nutrients. After eating, ghrelin abruptly declines, with levels varying 2- to 3-fold between the fasted and fed states. Interestingly, in obesity and type 2 diabetes (T2D), this pattern is disrupted. Individuals with these disorders have chronically suppressed ghrelin levels and little variation before and after meals.

Although ghrelin's preprandial rise and postprandial fall is a well-established phenomenon, its role in regulating glucose metabolism is unclear. In mice, increasing preprandial ghrelin levels improves glucose tolerance through enhanced glucagon-like peptide-1 (GLP-1) secretion. Ghrelin also stimulates GLP-1 secretion from mouse and human intestinal L-cells in vitro. These findings suggest enhanced postprandial GLP-1 as a novel role for the preprandial ghrelin surge. A ghrelin-incretin enteroendocrine axis could also explain the poor postprandial GLP-1 secretion and glucose tolerance in subjects with T2D, given their preprandial hypoghrelinemia.

The investigators' preliminary data demonstrate that in humans, increasing circulating ghrelin to a supraphysiologic range worsened glucose tolerance, despite increased GLP-1 secretion. The discrepancy between these findings and the ones from rodents could be due to difference in study design and/or species. For example, the investigators' study used a continuous ghrelin infusion, which resulted in elevated levels of ghrelin pre- and postprandially. Elevated postprandial ghrelin likely mitigated the positive effects of increased GLP-1 secretion by raising levels of glucagon and other counter-regulatory hormones.

This study seeks to delineate the interactions between ghrelin and GLP-1 in the regulation of glucose tolerance, beta-cell function, and insulin sensitivity. The investigators hypothesize that increased preprandial ghrelin will enhance GLP-1 secretion and consequently improve glucose tolerance in healthy subjects and those with T2D. Confirmation of these hypotheses would advance the investigators understanding of the control of glucose homeostasis and have important clinical and therapeutic implications. Modulating ghrelin levels may provide a novel therapeutic strategy to improve glucose tolerance in individuals with T2D, which affects an estimated 350 million people worldwide.

ELIGIBILITY:
Inclusion Criteria:

T2DM study subjects must meet the following inclusion criteria:

* established T2DM with good to moderate glycemic control (HbA1c ≤ 8.5%)
* Diabetes treated with oral medications or lifestyle management
* BMI 25.0 - 45.0 kg/m2

Healthy control subjects must meet the following inclusion criteria:

* Fasting glucose <100 mg/dL, as measured at screening visit
* HbA1c < 5.7%, as measured at screening visit
* BMI 18.0 - 29.9 kg/m2
* No diagnosis of diabetes mellitus (including gestational diabetes)
* Age between 18 - 40 years

Exclusion Criteria:

All subjects will be excluded for the following reasons:

* Active infections
* History of malignant or inflammatory conditions, such as rheumatoid arthritis and inflammatory bowel disease
* History of myocardial infarction or congestive heart failure
* History or active liver or renal disease (AST or ALT >2x upper limits of normal, calculated glomerular filtration rate [eGFR] <60 at screening)
* Anemia defined as hematocrit <34% at screening visit
* Uncontrolled hypertension
* History of pituitary or adrenal disorders or neuroendocrine tumor
* History of anorexia nervosa or previous gastrointestinal surgery
* Malabsorptive GI disease, such as celiac disease
* Pregnancy or lactation
* Use of medications that alter glucose metabolism or GI function (glucocorticoids, psychotropics, niacin, narcotic, metoclopramide)
* Use of insulin or GLP-1 based therapy (i.e. DPP-4 inhibitors, GLP-1 receptor agonists)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Effect of preprandial ghrelin on glucose tolerance | Approximately 4-8 weeks
  Primary Outcome: Glucose area under the curve during 60-minute Meal Tolerance test in healthy subjects and in Type 2 diabetic subjects

SECONDARY OUTCOMES:
Effect of preprandial ghrelin on GLP-1 secretion | Approx 4-8 weeks
  Secondary Outcome: Effect of preprandial ghrelin on GLP-1 area under the curve during a mixed meal in healthy subjects and in Type 2 diabetic subjects
Effect of preprandial ghrelin on insulin secretion | Approx 4-8 weeks
  Secondary Outcome: Effect of preprandial ghrelin on insulin and c-peptide area under the curve during a mixed meal in healthy subjects and in Type 2 diabetic subjects
Effect of preprandial ghrelin on beta cell function | Approx 4-8 weeks
  Secondary Outcome: Effect of preprandial ghrelin on beta cell function (as measured by Disposition Index = [ (Area under the insulin curve / Area under the glucose curve) X Matsuda Index] during a 60-minute Meal Tolerance test in healthy subjects and in Type 2 diabetic subjects
Effect of preprandial ghrelin on insulin sensitivity (as measured by Matsuda index) | Approx 4-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Tong, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center For Living, Durham, North Carolina, United States